CLINICAL TRIAL: NCT06120075
Title: A Phase 1/1b Study to Evaluate the Safety and Tolerability of AB801 Monotherapy and Combination Therapy in Participants With Advanced Malignancies
Brief Title: A Study of AB801 Monotherapy and Combination Therapy in Participants With Advanced Malignancies
Acronym: ARC-27
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-27
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancer
Keywords: AB801; Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation Cohort 1 - AB801 capsule Dose Level 1 (Experimental): Participants will receive AB801 orally daily
  Interventions: Drug: AB801
- Dose Escalation Cohort 2 - AB801 capsule Dose Level 2 (Experimental): Participants will receive AB801 orally daily
  Interventions: Drug: AB801
- Dose Escalation Cohort 3 - AB801 capsule Dose Level 3 (Experimental): Participants will receive AB801 orally daily
  Interventions: Drug: AB801
- Dose Escalation Cohort 4 - AB801 capsule Dose Level 4 (Experimental): Participants will receive AB801 orally daily
  Interventions: Drug: AB801
- Dose Escalation Cohort 5 - AB801 tablets Dose Level 5 (Experimental): Participants will receive AB801 orally daily
  Interventions: Drug: AB801
- Dose Escalation Cohort 6 - AB801 tablets Dose Level 6 (Experimental): Participants will receive AB801 orally daily
  Interventions: Drug: AB801
- Dose Escalation Cohort 7 - AB801 tablets Dose Level 7 (Experimental): Participants will receive AB801 orally daily
  Interventions: Drug: AB801
- Dose Expansion Cohort - AB801 + Docetaxel (Experimental): Participants with NSCLC will receive AB801 orally in combination with docetaxel IV infusion
  Interventions: Drug: AB801; Drug: Docetaxel

INTERVENTIONS:
Drug: AB801 — Administered as specified in the treatment arm
Drug: Docetaxel — Administered as specified in the treatment arm
  Arms: Dose Expansion Cohort - AB801 + Docetaxel

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AB801 in participants with advanced malignancies, and to determine a recommended AB801 dose for expansion.

ELIGIBILITY:
Key Inclusion Criteria:

* Monotherapy-specific criteria for dose escalation cohorts:

  * Participants may have cytologically or pathologically confirmed non-small cell lung carcinoma (NSCLC), colorectal carcinoma (CRC), breast, ovarian, renal cell carcinoma (RCC), head and neck squamous cell carcinoma (HNSCC), or bladder (including urothelial malignancies of the renal pelvis and ureter) carcinoma that has progressed or was non-responsive to available therapies with no standard of care (SOC) options, or for whom standard therapy has proven ineffective, intolerable, or considered inappropriate; or for whom a clinical study of an investigational agent is a recognized SOC.
* Disease-specific criteria for dose-expansion (NSCLC):

  * Cytologically or pathologically confirmed locally advanced unresectable or metastatic (Stage IIIB-IV per American Joint Committee on Cancer version 8) non-squamous NSCLC negative for actionable mutations in EGFR, ALK, ROS1, NTRK, C-MET, or RET. Mixed SCLC and squamous NSCLC histology is not permitted.
  * Previously treated in the unresectable locally advanced or metastatic setting with a platinum-containing chemotherapy and PD-(L)-1inhibitor.
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) guidance (Version 1.1) (Section 1.1). The measurable lesion must be outside of a radiation field if the participant received prior radiation unless discussed and approved by the study physician.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

Key Exclusion Criteria:

* Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of initiation of investigational product.
* Underlying medical conditions or adverse events that, in the physician or sponsor's opinion, will make the administration of investigational products hazardous.
* Prolonged QT interval defined as mean corrected QT interval (QTc) ≥ 450 milliseconds (ms).
* Any active or documented history of autoimmune disease, including but not limited to inflammatory bowel disease, celiac disease, Wegner syndrome, Hashimoto syndrome, systemic lupus erythematosus, scleroderma, sarcoidosis, or autoimmune hepatitis, within 3 years of the first dose of study treatment.
* Treatment with systemic immunosuppressive medication (including but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor-α agents) administered within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressant medication during study treatment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to 2 years
Dose Escalation Cohorts: Number of Participants With Dose-Limiting Toxicities (DLTs) | Up to 2 years

SECONDARY OUTCOMES:
Area Under the Plasma Drug Concentration-Time Curve (AUC) | Predose, Up to 8 hours postdose
Maximum Concentration (Cmax) in Plasma | Predose, Up to 8 hours postdose
Time to Maximum Concentration (Tmax) in Plasma | Predose, Up to 8 hours postdose
Objective response rate (ORR) as Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 2 years
Dose Expansion Cohorts: Duration of Response (DOR) as Assessed per RECIST v1.1 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (10):
- United States (10):
  - Sarah Cannon Research Institute, Denver, Colorado
  - Georgetown, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - START Midwest, Grand Rapids, Michigan
  - Icahn School of Medicine at Mount Sinai/ The Tisch Cancer Center, New York, New York
  - University Of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley, Dallas, Texas
  - START - South Texas Accelerated Research Therapeutics, LLC., San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Next Oncology Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-27 - Public website — https://trials.arcusbio.com/study/?id=ARC-27